CLINICAL TRIAL: NCT05187572
Title: Effectiveness of Reminiscence Therapy Versus Cognitive Stimulation in Older Adults With Cognitive Decline: a Quasi-experimental Pilot Study
Brief Title: Effectiveness of Reminiscence Therapy Versus Cognitive Stimulation in Older Adults With Cognitive Decline
Acronym: TRvsCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulo Costa (Other)
Collaborators: Junta de Freguesia de Santo António dos Olivais (Unknown); Centro Sociocultural Polivalente de São Martinho (Unknown); Centro Social e Paroquial de Carapinheira do Campo (Unknown); Obra Social de Torre de Vilela (Unknown); Centro Social Paroquial de Pedrulha (Unknown); Associação Nacional de Apoio ao Idoso (Unknown); Santa Casa de Misericórdia de Cantanhede (Unknown); Doce Viver - Residencial Sénior, Bruscos (Unknown)
Responsible Party: Sponsor-Investigator, Paulo Costa, Researcher, Escola Superior de Enfermagem de Coimbra
Organization: Escola Superior de Enfermagem de Coimbra (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TRvsCS
Record Dates: First submitted 2021-12-21; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Treatment allocation will be done per institution, after a centralized randomization process. Care providers and outcome assessors will be blinded to the allocation process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminiscence Therapy (RT) (Experimental): The RT program is composed of activities that follow older adults' lifespan (e.g., school, professional life, travelling, holidays and celebrations, historical dates/moments). Such activities allow older adults to revive and share life-changing/significant moments and integrate them into their autobiographical narrative. The program was developed and validated by Gil and colleagues for Portuguese older adults with cognitive decline.
  Interventions: Behavioral: Group intervention
- Cognitive Stimulation (CST) (Experimental): The CST intervention was based on the "Making a Difference" program, specifically developed for older adults with cognitive decline and previously adapted and validated to the European Portuguese language and culture. This program offers a sequence of activities that covers different cognitive domains and promotes older adults' socialization and self-esteem.
  Interventions: Behavioral: Group intervention

INTERVENTIONS:
Behavioral: Group intervention — This intervention was developed during 14 sessions, held twice a week, with a duration of 45 to 60 minutes each. The sessions were developed as group-based interventions, facilitated by a leader and a co-leader from each community institution.

SUMMARY:
Although data suggest that non-pharmacologic therapies such as Reminiscence Therapy (RT) and Cognitive Stimulation (CS) can potentially maintain or reverse this trend, cognitive impairment can be a precursor to neurodegenerative processes. This study aimed to assess how an RT and a CS program affected cognition, depressive symptomatology, and quality of life (QoL) in older persons with cognitive decline who attended community support institutions in central Portugal. For seven weeks, a quasi-experimental study with two arms (RT and CS program) was conducted. The intervention was completed by 76 of the 109 older persons who were first screened (50 in the RT program, 26 in the CS program). In both groups, a pre- and post-intervention analysis revealed statistically significant differences in cognition, particularly in older adults' delayed recall ability.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent before study commencement;
* Ability to participate in group activities for a period between 45 to 60 minutes;
* No pronounced impairment of their visual and auditory abilities;
* Mild to moderate cognitive decline, assessed as a score equal to or below 20 points in the Six-Item Cognitive Impairment Test (6-CIT).

Exclusion Criteria:

* Unstable clinical condition;
* Prescribed with cholinesterase inhibitors and/or antipsychotics during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Change in cognition (person with cognitive decline) | Pre-intervention (baseline)
  Measured using the Montreal Cognitive Assessment (MoCA). Scale scores vary between 0 and 30 points; higher scores correspond to a higher cognition level.
Change in depressive dymptomatology (person with cognitive decline) | Pre-intervention (baseline)
  Measured using the 10-items Geriatric Depression Scale (GDS-10). Scale scores vary between 0 and 10 points; scores equal or above 2 points correspond to a screening diagnosis of depression.
Change in quality of life (person with cognitive decline) | Pre-intervention (baseline)
  Measured using the World Health Organization Quality of Life - module for older adults (WHOQOL-OLD-8). Scale scores vary between 8 and 40 points; higher scores correspond to a higher level of quality of life.
Change in cognition (person with cognitive decline) | 8 weeks post baseline
  Measured using the Montreal Cognitive Assessment (MoCA). Scale scores vary between 0 and 30 points; higher scores correspond to a higher cognition level.
Change in depressive dymptomatology (person with cognitive decline) | 8 weeks post baseline
  Measured using the 10-items Geriatric Depression Scale (GDS-10). Scale scores vary between 0 and 10 points; scores equal or above 2 points correspond to a screening diagnosis of depression.
Change in quality of life (person with cognitive decline) | Pre-intervention (baseline), 8 weeks post baseline
  Measured using the World Health Organization Quality of Life - module for older adults (WHOQOL-OLD-8). Scale scores vary between 8 and 40 points; higher scores correspond to a higher level of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Silva, PhD, Study Chair — Health Sciences Research Unit: Nursing, Nursing School of Coimbra; João Apóstolo, PhD, Study Director — Health Sciences Research Unit: Nursing, Nursing School of Coimbra
Locations (1):
- The Health Sciences Research Unit: Nursing, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available on request. The data are not publicly available due to ethical considerations, regarding personal information and respecting what was written in the signed informed consent.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data presented in this study are available on request. The data are not publicly available due to ethical considerations, regarding personal information and respecting what was written in the signed informed consent.
Access Criteria: The data presented in this study are available on request. The data are not publicly available due to ethical considerations, regarding personal information and respecting what was written in the signed informed consent.

REFERENCES:
- See also: Project website — http://www.esenfc.pt/ecog